CLINICAL TRIAL: NCT03387449
Title: Adaptive Arm Training for Children With Hemiplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Blythedale Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BAT_Friel
Record Dates: First submitted 2017-12-22; First posted 2018-01-02 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2022-01

CONDITIONS: Cerebral Palsy; Hemiplegia; Hemiparesis; Acquired Brain Injury
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia; Paresis; Brain Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Bimanual Arm Training (Experimental): Children in the study will all receive the same treatment, which includes 9 weeks of training on the bimanual arm trainer robotic device.
  Interventions: Device: Bimanual Arm Training

INTERVENTIONS:
Device: Bimanual Arm Training — Device-based bimanual-to-unimanual training will be provided with the Bimanual Arm Trainer (BAT, Mirrored Motion Works, NC). The device provides bimanual-to-unimanual training of simultaneous shoulder external rotation and elbow extension, and independent training of pronation-supination and grasp and release of each hand. Range of motion and speed are recorded during training and feedback and motivation are provided through age-appropriate gaming modules.

SUMMARY:
The goal of this research is to provide limb training in children with hemiplegia using a bimanual-to-unimanual training approach. Twenty pediatric patients aged 5-17 years with acquired brain injury will receive training on the bimanual-to-unimanual device for a period of 9 weeks. During the training, children use both arms to operate robotic arms to play a video game. We will assess changes in hand impairment after the training.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegia due to brain injury at least 3 months before study enrollment.

Exclusion Criteria:

* Any social or medical problem that precludes compliance with the protocol.
* Treatment with botulinum toxin or intrathecal baclofen in the 3 months preceding enrollment.
* Implanted neuromodulatory or electronic device or other complicating illness.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2017-11-07 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in Assisting Hand Assessment | Before intervention compared to after intervention
  The Assisting Hand Assessment evaluated how effectively children use their hands to complete bimanual tasks.
Change in Box and Box Test | Before intervention compared to after intervention
  The Box and Blocks test measures how many blocks a child can move with one hand from one box to another in one minute with the impaired hand.
Change in range of motion | Before intervention compared to after intervention
  The robotic device measures range of motion of the shoulder.

CONTACTS AND LOCATIONS:
Locations (1):
- Kathleen M Friel, Hartsdale, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
We plan to share results with our collaborator Dr. Preeti Raghaven, at New York University. Dr. Raghavan created the robot we are using, has IRB approval to use the robot, and is a consultant on this study. Personal health information will not be shared.
Supporting Information: Study Protocol, SAP
Time Frame: during the study